CLINICAL TRIAL: NCT05132907
Title: Phase 1, Dose-Escalation Study of Nanoparticle Carrier-Formulated Self- Replicating Replicon RNA (repRNA) SARS-CoV-2 Vaccine (HDT-301) Targeting a Variant Spike Protein in Unvaccinated or Previously Vaccinated Healthy Adults
Brief Title: Safety and Immunogenicity of HDT-301 Targeting a SARS-CoV-2 Variant Spike Protein
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HDT Bio (Industry)
Collaborators: Rainier Clinical Research Center (Other); C3 Research Associates (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HDT-301-002
Record Dates: First submitted 2021-11-18; First posted 2021-11-24 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: SARS-CoV2 Infection
MeSH Terms: conditions — COVID-19 | interventions — repRNA-CoV2S vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1 (previously vaccinated, two dose recipients) (Experimental): Cohort 1 will include individuals with vaccination against COVID-19 who will receive a two-dose schedule of HDT-301 56 days apart. Dose will be escalated from low to mid to high according to predefined safety parameters.
  Interventions: Biological: HDT-301
- Cohort 2 (previously vaccinated, single dose recipients) (Experimental): Cohort 2 will include individuals with vaccination against COVID-19 who will receive a one-dose schedule of HDT-301. Dose will be escalated from low to mid to high according to predefined safety parameters.
  Interventions: Biological: HDT-301
- Cohort 3 (previously unvaccinated) (Experimental): Cohort 3 will include 21 individuals with no history of vaccination against COVID-19 who will receive a two-dose schedule of HDT-301 56 days apart. Dose will be escalated from low to mid to high according to predefined safety parameters.
  Interventions: Biological: HDT-301

INTERVENTIONS:
Biological: HDT-301 — HDT-301 Investigational Vaccine (a Nanoparticle Carrier-Formulated Replicon RNA (repRNA-CoV2S))

SUMMARY:
This is Phase 1 study is to assess tolerability and immunogenicity of three dose levels of the investigational HDT-301 vaccine administered intramuscularly (IM), both in immunization-naïve participants and as a booster for those participants who previously received a SARS-CoV-2 vaccine.

Safety and tolerability will be the primary endpoint assessed by incidence of adverse events at each dose through 12 months after completion of the vaccination regimen (either one dose, or two doses provided 56 days apart). Immunogenicity evaluations will be conducted for pre-specified timepoints as secondary and exploratory endpoints.

DETAILED DESCRIPTION:
This is an open-label, dose-ranging, study to evaluate the safety and immunogenicity of the investigational HDT-301 vaccine in healthy (vaccinated or unvaccinated) adult subjects, with a 4:3 recruitment of individual aged 18-49 years and 50-65 years, respectively. The study duration is approximately 13 or 14 months for each subject.

Three cohorts of 21 subjects each will be sequentially recruited in the study:

1. Cohort 1 will include individuals with vaccination against COVID-19 who will receive a two-dose schedule of HDT-301 56 days apart.
2. Cohort 2 will include individuals with vaccination against COVID-19 who will receive a one-dose schedule of HDT-301.
3. Cohort 3 will include individuals with no history of vaccination against COVID-19 who will receive a two-dose schedule of HDT-301 56 days apart.

Recruiting and screening of participants will be conducted on a continual basis. Subjects confirmed to be Emergency Use Authorization (EUA) SARS-CoV-2 vaccine recipients will first be placed into either Cohort 1 (Study Days 1 and 57; Two-Dose Regimen) or Cohort 2 (Study Day 1; One-Dose Regimen) then subsequently placed into each of the three dose groups. Subjects in the Cohort 3 (naïve, unimmunized) subset will be placed into each of the three dose groups to receive the study vaccine on Study Days 1 and 57 (Two-Dose Regimen). Each cohort will be divided into 3 groups of 7 participants, that will be provided HDT-301 at either a low-, mid- or high-dose. For each of the three-dose groups, a sentinel group will be initially enrolled and followed through Day 8 post-dose one for safety. If no halting rules are met by Day 8 enrollment will proceed to the remaining subjects. Blood samples will be collected during the study for each participant.

ELIGIBILITY:
Inclusion Criteria:

-

Each subject must meet ALL of the following criteria in order to participate in this study:

1. Male or non-pregnant female 18 through 65 years of age at the time of first vaccination.
2. Known clinical and immunization status versus SARS-CoV-2.

   1. For Cohort 3 participants this will be either no history of COVID-19 nor reported history of vaccination against COVID-19 by Emergency Use Authorization (EUA) vaccine or investigational product.
   2. For Cohort 1 and Cohort 2 participants, this will be verified receipt of investigational or Emergency Use Authorization (EUA) vaccines against SARS-CoV-2 (by provision of either access to medical records, Washington state online vaccine registry, documentation of receipt of investigational vaccine, or Vaccine Card), with most recent vaccination 90 days or more prior to trial initiation (days of immunization will be noted, along with vaccine manufacturer).
3. Understands and agrees to comply with the study procedures and provides written informed consent.
4. In the opinion of the PI or designee, could and would comply with the requirements of the protocol (e.g., completion of Memory Aids, return for follow-up visits, availability for safety calls).
5. Body mass index ≥18.0 and ≤35.0 kg/m2.
6. Considered by the PI or designee to be in good general health as determined by medical history, clinical laboratory assessments, vital sign measurements, and physical examination findings at Screening.
7. Women of childbearing potential1 must agree to use or have practiced true abstinence or use at least one acceptable primary form of contraception. These criteria are applicable to females in a heterosexual relationship and of childbearing potential (i.e., the criteria do not apply to subjects in a same sex relationship).
8. Female subjects of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test on the day of and prior to each study vaccination.
9. Must agree to refrain from donating blood or plasma during the study (outside of this study).

Exclusion Criteria:

-

To participate in this study, all subjects must meet NONE of the exclusion criteria described:

1. Female subject who is breastfeeding or plans to breastfeed from the time of the first vaccination through 60 days after the last vaccination.
2. Has any medical disease or condition that, in the opinion of the participating site PI or appropriate sub-investigator, precludes study participation.
3. Presence of self-reported or medically documented significant medical or psychiatric condition(s).
4. History of hypersensitivity or severe reactions to previous vaccinations (e.g., anaphylaxis, urticaria, other significant reaction requiring medical intervention).
5. History of hypersensitivity or severe reactions to products known to contain polyethylene glycol (PEG).
6. Subjects with a positive test result at Screening for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus types 1 or 2 antibodies.
7. Known or suspected alcohol or drug abuse within the past 6 months prior to Screening.
8. Safety laboratory test results (hematology and chemistry) with a toxicity score ≥ Grade 2 at Screening. The inclusion of subjects with non-clinically significant (NCS) Grade 1 laboratory or vital sign abnormalities is allowed based on investigator's discretion (e.g., oral temperature is less than 100.0°F (37.8°C); pulse no greater than 100 beats per minute; systolic BP is 85 to 150 mm Hg, inclusive).
9. Previous participation in other studies involving study intervention containing lipid nanoparticles.
10. Clinical conditions representing a contraindication to intramuscular vaccination and blood draws.
11. Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs within 6 months prior to the first vaccine dose (for corticosteroids: prednisone ≥ 20 mg/day or equivalent). Inhaled, nasal and topical steroids are allowed.
12. Received immunoglobulins or any blood products within 3 months prior to any study vaccination.
13. Received an investigational or non-registered medicinal product within 30 days prior to informed consent.
14. Has any blood dyscrasias or significant disorder of coagulation.
15. Has any chronic liver disease, including fatty liver.
16. Received or plans to receive a licensed, live vaccine within 4 weeks before or after each vaccination.
17. Received or plans to receive a licensed, inactivated vaccine within 2 weeks before or after each vaccination.
18. Has an acute illness, as determined by the participating site PI or appropriate sub- investigator, with or without fever (oral temperature ≥38.0°C [100.4°F]) within 72 hours prior to each vaccination.
19. Any medical, psychiatric, or occupational condition which, in the opinion of the investigator, might pose additional risk to the subject due to participation in the study or could interfere with evaluation of the study vaccine or interpretation of study results.
20. Unknown vaccine status versus SARS-CoV-2.
21. Receipt of Emergency Use Authorization or other vaccines against SARS-CoV-2 infection within 90 days prior to administration of first dose (recruits in Cohort 3 will be unimmunized; recruits in Cohorts 1 and 2 will have completed their Emergency Use Authorization (EUA) vaccine regimen at least 90 days prior to enrolment).
22. Regular smoking or vaping (more than three days per week).
23. Study personnel or immediate family or household member of study personnel.
24. The subject has donated blood within 56 days of dosing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Solicited AE | Day 1-71
  Frequency and grade of solicited local and systemic AEs during a 14 day follow-up period after each vaccination (i.e., the day of vaccination and 14 subsequent days).
Unsolicited AE | Day 1-85
  Frequency and grade of any unsolicited AE within a 28 day period following each vaccination (i.e., the day of vaccination and 28 subsequent days).
Lab abnormalities | Day 1-85
  Occurrence of any laboratory abnormality (increased or decreased outside normal ranges, as determined by toxicity scales) at 7 and 28 days after each vaccination.
Medically-attended AE, AESI and SAE | Day 1-422
  Occurrence of medically-attended AEs and NOCMCs during the entire study period. Occurrence of AESIs during the entire study period. Occurrence of SAEs during the entire study period.

SECONDARY OUTCOMES:
Immunogenicity Endpoints (magnitude of IgG response) | Day 1-85
  Geometric Mean Titer (GMT) of SARS-CoV-2 B.1.351 Spike-specific IgG by ELISA 28 days after the first (or only) vaccination (Study Day 29) and 28 days after the second vaccination (Study Day 85).
Immunogenicity Endpoints (proportion of IgG responders) | Day 1-85
  Proportion of subjects with a ≥4-fold increase in SARS-CoV-2 B.1.351 Spike-antibody titer from baseline to 28 days after the first (or only) vaccination (Study Day 29) and at 28 days after the second vaccination (Study Day 85), determined by a validated SARS-CoV-2 specific IgG by ELISA.
Immunogenicity Endpoints (magnitude of neutralizing antibodies) | Day 1-85
  Geometric mean titer (GMT) of SARS-CoV-2 B.1.351-specific serum neutralizing antibodies 28 days after the first (or only) vaccination (Study Day 29) and 28 days after the second vaccination (Study Day 85).
Immunogenicity Endpoints (proportion responding with neutralizing antibodies) | Day 1-85
  Proportion of subjects with a ≥4-fold increase in SARS-CoV-2 B.1.351-specific serum neutralizing antibody titers from baseline to 28 days after the first (or only) vaccination (Study Day 29; and at 28 days after the second vaccination (Study Day 85).

OTHER OUTCOMES:
Exploratory Immunology (IgG isotype profile and magnitude) | Day 1-422
  Geometric mean titer (GMT) of SARS-CoV-2 B.1.351 Spike-specific IgG1, IgG2, IgG3, and IgG4 by ELISA.
Exploratory Immunology (proportion with IgG isotype profile) | Day 1-422
  Proportion of subjects with a ≥ 4-fold increase in SARS-CoV-2 B.1.351 Spike-specific IgG1, IgG2, IgG3, and IgG4 ELISA antibody titers from baseline to post-vaccination time points.
Exploratory Immunology (magnitude alternate antibodies) | Day 1-422
  Geometric mean titer (GMT) of SARS-CoV-2 B.1.351 Spike-specific IgM and IgA by ELISA.
Exploratory Immunology (proportion with alternate antibodies) | Day 1-422
  Proportion of subjects with a ≥ 4-fold increase in SARS-CoV-2 B.1.351 Spike-specific IgM and IgA antibody titers from baseline to post-vaccination time points.
Exploratory Immunology (response against heterologous Spike) | Day 1-422
  Geometric mean titer (GMT) of IgG binding SARS-CoV-2 Spike of genetic sequences distinct from the vaccine B.1.351 Spike sequence.
Exploratory Immunology (T cell phenotype) | Day 1-422
  Diversity of the T cell responses by assessing cells expressing interferon gamma (IFN-γ), interleukin 2 (IL-2), tumor necrosis factor (TNF), and other markers.

CONTACTS AND LOCATIONS:
Overall Officials: Steven G Reed, Ph.D, Principal Investigator — HDT Bio
Locations (1):
- Rainier Clinical Research, Renton, Washington, United States

IPD SHARING:
Plan to Share IPD: No